CLINICAL TRIAL: NCT03930056
Title: Micro-Processor Controlled Knee-Ankle-Foot Orthosis (C-Brace) Usage in a Spinal Cord Injury (SCI) Population Compared to Traditional Rehabilitation Methods: Determining Functional Outcome Differences of Recovery
Brief Title: C-Brace II Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00208781
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury
Keywords: Orthotic; C-Brace
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- C-Brace II Group (Experimental): Subjects will be assigned a C-Brace II orthotic for use.
  Interventions: Device: C-Brace II
- Traditional Group (Active Comparator): Subjects will continue with their own KAFO (non C-Brace II) use.
  Interventions: Device: Traditional Care KAFO intervention

INTERVENTIONS:
Device: C-Brace II — Participant will complete 3-6 orthoses sessions to complete clinical evaluations and fittings conducted by certified orthotists.
  Participant will receive 10-20, one hour training sessions over 1-2 months in the lab. These sessions include tuning the device and system tweaks in accordance to needs/preferences of participant, vitals signs, skin checks, pain, and exertion levels. Sessions involve training with the device, which includes putting on / taking off the device, transfer training, gait training, and balance and fall prevention.
  Up to 20 sessions will be conducted until minimum safety guidelines are reached during a minimum of at least 3 training sessions in a row.
  Participant will take the assigned device home to use for a 3-month period. Participant will be given an activity monitor to wear at all times except showering and instructed how to charge the device and use it. Participant will return for testing at 3, 6 and 12 months after receiving the brace for testing.
  Arms: C-Brace II Group
Device: Traditional Care KAFO intervention — Participant will continue with use of their own KAFO. Participant will receive 10-20, one hour training sessions over 1-2 months in the lab, if Patient is not already receiving care in a therapy setting. These sessions include tuning the device and system tweaks in accordance to needs/preferences of participant, vitals signs, skin checks, pain, and exertion levels. Sessions involve training with the device, which includes putting on / taking off the device, transfer training, gait training, and balance and fall prevention. Up to 20 sessions will be conducted until minimum safety guidelines are reached during a minimum of at least 3 training sessions in a row. Participant will continue with the assigned device home to use for a 3-month period. Participant will be given an activity monitor to wear at all times except showering and instructed how to charge the device and use it. Participant will return for testing at 3, 6 and 12 months after receiving the brace for testing.
  Arms: Traditional Group

SUMMARY:
A randomized, repeated measures comparative design study to compare use of a micro-processor controlled knee-ankle-foot orthosis vs. traditional care knee-ankle-foot-orthosis (KAFO) models following discharge from inpatient rehabilitation.

ELIGIBILITY:
All participants:

Inclusion Criteria:

* Be within 3-24 months post spinal cord injury diagnosis
* 18-80 years
* Must be able to demonstrate the ability to charge assigned sensors during 3-month home trial period on and off and sufficient memory ability to wear the devices each day during use of the orthoses.

Exclusion Criteria:

* Unstable neurological, cardiovascular, or cancer diagnoses.
* Cognitive impairments that limit study participation

In addition to the above inclusion criteria, the following criteria must be met to be designated into the study interventional tract (C-Brace II):

Inclusion criteria:

* Requires orthotic bracing for lower extremity instability, including the knee joint, unilaterally or bilaterally

Exclusion criteria:

* Body weight over 275 lbs
* Flexion contracture in the knee and/or hip joint in excess of 10 degrees
* Non-correctable knee varus/valgus in excess of 10 degrees
* Moderate to severe spasticity
* Leg length discrepancy in excess of 6" (15.24 cm)
* Inability to stabilize the trunk with or without assistive devices (crutches, cane, etc.)
* Inability to successfully use C-Brace trial tool in advancement of leg/s.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk Test (6MWT) | Change from baseline in 6MWT distance after using device at 3, 6, and 12 month follow-up.
  The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption.

SECONDARY OUTCOMES:
Muscle Strength (manual muscle test) | Change from baseline in muscle strength after using device at 3, 6, and 12 month follow-up.
  Muscle strength will be assessed by a trained clinical researcher
Passive and Active Range of Motion of Lower Extremity joints | Change from baseline in range of motion after using device at 3, 6, and 12 month follow-up.
Modified Ashworth Scale | Change from baseline in muscle tone after using device at 3, 6, and 12 month follow-up.
  A scale used to measure the amount of tone in individuals with neurologic diagnoses. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
10 Meter Walk Test (10MWT) | Change from baseline in gait speed after using device at 3, 6, and 12 month follow-up.
  This test will examine the patient's gait speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire 10 meter distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundred of a second (ex: 2.15 sec). The test will be recorded 6 times: 3 times at the patient's self-selected speed, and 3 times at the patient's quickest, yet safest speed. The average of each of the 3 times will be recorded. Adequate rest in between trials will be given.
Walking Index for Spinal Cord Injury (WISCI II) | Change from baseline in rank score after using device at 3, 6, and 12 month follow-up.
  A rank ordering along a dimension of impairment, from the level of most severe impairment (0) to least severe impairment (20) based on the use of devices, braces, and physical assistance of one or more persons.
Functional Gait Assessment (FGA) | Change from baseline in FGA score after using device at 3, 6, and 12 month follow-up.
  The Functional Gait Assessment is a 10 item test used to assess postural stability during walking tasks. It has a maximum score of 30 with each item being scored 0-3. It may be performed with or without an assistive device; however, individuals lose a point on all items requiring a device.
Berg Balance Scale (BBS) | Change from baseline in Berg Balance score after using device at 3, 6, and 12 month follow-up.
  The Berg Balance Scale is a 14-item scale designed to measure balance in adults in a clinical setting. When scoring, the lowest response category that applies should be recorded. In each item, points should be deducted if the time or distance requirements are not met, the subject's performance requires supervision, or the subject requires assistance from support or examiner.
Timed Up and Go test (TUG) | Change from baseline in TUG score after using device at 3, 6, and 12 month follow-up.
  A test which times the ability of a patient to stand up from a standard chair with arm rests, walk 3 meters forward, turn around, walk 3 meters back to the chair, and sit back down in the chair.
Gaitrite data capture | Change from baseline in gait parameters after using device at 3, 6, and 12 month follow-up.
  The Gaitrite system automates measuring temporal and spatial gait parameters via an electronic walkway connected to a computer. The Gaitrite electronic walkway contains sensor pads encapsulated in a carpet to collect gait information. The system can be laid over any flat surface. The Gaitrite electronic walkway for the study shall be a minimum of 14 feet long. The Gaitrite data capture was chosen as measurement of the patient's overall gait quality. Patients will be asked to walk at a self-selected speed across the Gaitrite electronic walkway.

OTHER OUTCOMES:
Activities Specific Balance Confidence Scale (ABC) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The ABC Scale is a self-report questionnaire consisting of 16 items designed to measure fear of falling. It assesses an individual's perception of balance during activities of daily living by asking the individual to rate their confidence during different activities on a 0% (no confidence) to 100% (completely confident) scale.
Modified Falls Efficacy Scale (mFES) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling."
Spinal Cord Injury Quality of Life (SCI-QOL) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The SCI-QOL are a battery of self-reported questionnaires completed by participants to evaluate perceptions of personal independence, ability to communicate needs with others, and sense of control over one's life in individuals with spinal cord injury.
EQ5D-5L | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  A self-reported, health related, quality of life questionnaire. It measures quality of life in 5-components including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on a scale describing the degree of problems in that area. It ends with an overall health scale between 1-100 to rate the level of health the user is experiencing at the time of the test.
Orthotics and Prosthetics User Survey (OPUS) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The Orthotic and prosthetics User Survey is a self-report questionnaire which is designed to evaluate the outcome of orthotic and prosthetic services. We will administer three of the five domains: lower limb functional measure, health-related quality of life, and satisfaction with device. The domains of upper limb functional measure and satisfaction with service are not applicable in this study.
World Health Organization Quality of Life (WHOQOL-BREF) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The WHOQOL-BREF is a self-report questionnaire that measures an individual's perceived quality of life. It contains four domains which cover physical health, psychological health, social relationships, and environment. Scores range from 0-100 with 100 indicating a higher quality of life. The scores can be broken down by domain or taken as a whole. The WHOQOL-BREF is valid cross-culturally.
International Spinal Cord Injury Bowel Function Data Set | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The purpose of this test is to standardize collection and reporting on the bowel in individuals with spinal cord injury. Questions include bowel care procedures, surgical procedures, time, frequency, and method of bowel practices.
International Spinal Cord Injury Lower urinary Tract Basic Data Set | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  The purpose of this test is to standardize collection and reporting of information on the lower urinary tract in individuals with spinal cord injury. Questions include surgical procedures, drugs, bladder emptying, and incontinence. These are used by clinicians and researchers so that data can be shared and combined easily.
Spinal Cord Injury Bowel and Bladder Treatment Index Short Form (SCI-BBTI-SF) | Change from baseline in score after using device at 3, 6, and 12 month follow-up.
  A self-report questionnaire that assesses bowel and bladder function. It includes items regarding bowel and bladder emptying habit, complications from SCI-related surgery, assistance required, and perceived quality of life.
Actigraph | Change from baseline measurement after using device at 3, 6, and 12 month follow-up.
  The Actigraph is a small accelerometer worn on a body part which can identify performance of functional activities during use.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States